CLINICAL TRIAL: NCT00076492
Title: A Multi-center, Double-blind, Pilot Study of CoQ10 and GPI 1485 in Subjects With Early Untreated Parkinson's Disease
Brief Title: NINDS Parkinson's Disease Neuroprotection Trial of CoQ10 and GPI 1485
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Karl Kieburtz, Principal Investigator, University of Rochester
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: U01NS43128-2; U01NS043128 (NIH)
Record Dates: First submitted 2004-01-23; First posted 2004-01-27 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Parkinson disease; CoQ10; GPI 1485
MeSH Terms: conditions — Parkinson Disease | interventions — coenzyme Q10; GPI 1485

INTERVENTIONS:
Drug: CoQ10
Drug: GPI 1485

SUMMARY:
The goal of this study is to assess the impact of CoQ10 and GPI 1485 on the progression of Parkinson's disease, in order to determine whether it is reasonable to proceed with further study of either of these agents.

DETAILED DESCRIPTION:
Parkinson's disease (PD) affects nearly a million Americans, a number that will increase over the coming decades as the population ages. While available medical therapies are usually effective for controlling symptoms in the initial years following diagnosis, higher doses of multiple agents are required over time, with increasing side effects and incomplete control of symptoms. Although these treatments can dramatically improve the lives of patients with PD initially, they do not address the underlying causes of the disease or the inevitable disease progression.

This multi-center, randomized, double-blind trial will involve 42 trial centers in the United States and Canada, and enroll 195 people with PD. The primary objective of this neuroprotection trial is to identify agents capable of slowing the progression of PD. In the trial, investigators will assess the impact of CoQ10, an antioxidant, and GPI 1485, a novel immunophilin compound, on the progression of PD and determine if it is futile or non-futile to proceed with further study of these agents.

In this study, subjects with early, untreated PD will be equally randomized into one of the three study arms: 1.) the group that receives active CoQ10 and placebo instead of GPI 1485; 2.) the group that receives active GPI 1485 and placebo instead of CoQ10; or 3.) the group that receives placebo instead of CoQ10 and GPI 1485. Subjects will remain on the blinded study drug for 12 months.

ELIGIBILITY:
Inclusion:

* Willing and able to give informed consent.
* Men and women with idiopathic PD of less than 5 years duration from diagnosis.
* Diagnosis must be confirmed by bradykinesia plus one of the other cardinal signs (resting tremor, rigidity) being present, without any other known or suspected cause of parkinsonism. The clinical signs must be asymmetric.
* Subjects must not require any therapy (including levodopa, dopamine agonists, anticholinergics, amantadine, or selegiline) to treat symptoms of PD at the time of enrollment. Subjects may have had prior exposure to any one of these agents, but exposure with any agent may not have been longer than 60 days in duration and subjects must not have been on any of these agents within 90 days prior to baseline. Once a subject needs dopaminergic treatment, these medications may be added as part of best medical management. The subject will still remain in the study.
* Age > 30 years.
* Willingness and ability to comply with study requirements.
* Women who are not postmenopausal or surgically sterile must use a medically accepted contraceptive regimen for at least 60 days before the baseline visit, and agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug. Reliable forms of contraception include oral, implanted, or injected contraceptives; intrauterine devices in place for at least 3 months; or adequate barrier methods in conjunction with spermicide (abstinence is considered an acceptable contraceptive regimen). Women must have a pregnancy test unless they are at least 2 years postmenopausal or surgically sterile.

Exclusion:

* Use of any of the following drugs within 180 days prior to baseline: neuroleptics, metoclopramide, alpha-methyldopa, clozapine, olanzepine, and flunarizine.
* Use of any of the following drugs within 90 days prior to baseline: methylphenidate, cinnarizine, reserpine, amphetamine, or MAO-A inhibitors (pargyline, phenelzine, and tranylcypromine).
* Presence of atypical Parkinson's syndromes due to drugs (e.g., metoclopramide, flunarazine), metabolic identified neurogenetic disorders (e.g., Wilson's disease), encephalitis, or other degenerative diseases (e.g., progressive supranuclear palsy).
* Use of CoQ10 or GPI 1485 90 days prior to baseline.
* Use of minocycline or creatine 90 days prior to baseline.
* Receipt of other investigational drugs within 90 days prior to baseline.
* Presence of freezing.
* Impairment of postural reflexes (pull test score > 0).
* Any clinically significant medical condition (e.g., active GI illness, angina, active neoplasm) or laboratory abnormality, which would in the judgment of the investigator interfere with the subjects ability to participate in the study or to be followed.
* History of stereotaxic brain surgery for PD (e.g., pallidotomy, deep brain stimulation, fetal tissue implantation).
* Clinically significant structural brain disease that the investigator believes would interfere with study evaluations.
* Significant psychiatric disorders that may interfere with complying with the protocol.
* History of known hypersensitivity or intolerability to CoQ10 or GPI 1485.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195
Dates: Start 2004-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Kieburtz, MD, MPH, Principal Investigator — University of Rochester; Barbara Tilley, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Parashos SA, Luo S, Biglan KM, Bodis-Wollner I, He B, Liang GS, Ross GW, Tilley BC, Shulman LM; NET-PD Investigators. Measuring disease progression in early Parkinson disease: the National Institutes of Health Exploratory Trials in Parkinson Disease (NET-PD) experience. JAMA Neurol. 2014 Jun;71(6):710-6. doi: 10.1001/jamaneurol.2014.391. PMID 24711047